CLINICAL TRIAL: NCT02028923
Title: Phase III Study Evaluating the Efficacy of Topical Morphine in the Treatment of Severe Local Pain of Chronic Wounds
Brief Title: Efficacy of Topical Morphine in the Treatment of Severe Local Pain of Chronic Wounds
Acronym: EMGEL
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruiting patients too low
Sponsor: Institut Curie (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other); Hôpital Louis Mourier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IC 2013-01
Record Dates: First submitted 2014-01-06; First posted 2014-01-07 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-07

CONDITIONS: Local Pain; Chronic Wounds
Keywords: topical morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Morphine gel (Experimental): morphine 30 mg, quantity of gel per application: 15mg (15ml)
  Interventions: Drug: Morphine gel
- Neutral gel (Placebo Comparator): water for injection, quantity of gel per application: 15mg (15ml)
  Interventions: Other: Neutral gel

INTERVENTIONS:
Drug: Morphine gel — Topical
  Arms: Morphine gel
Other: Neutral gel — Topical
  Arms: Neutral gel

SUMMARY:
This phase III study aims to show that topical morphine low doses treats localized pain in chronic wounds, intense and rebellious to systemic analgesics included or not opioids.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged over 18 years
* Painful chronic wounds (bedsores, wound tumor, arterial ulcers, venous or mixed diabetic ulcer if systolic pressure index >0.8, necrotic angiodermatitis not graftable), a bottom surface 300 cm² and does not require more than 15 ml of gel by application. When patient has multiple painful chronic wounds, the wound having only the highest pain intensity is considered for evaluation.
* Ineffective systemic analgesic with or without opioid analgesic established and maintained at the same dose for 3 days before inclusion. If treatment includes morphine, the daily dose should not exceed 60 mg of morphine equivalent and this treatment must be a treatment exclusive background.
* Patient requiring an analgesic equilibration for intense and rebellious local pain, with a daily average score greater than or equal to 5, on a graduated numerical scale of 0 to 10. The score is defined at the inclusion and corresponds to the pain intensity felt locally by the patient under treatment systemic analgesic with or without co-analgesics.
* If analgesics to treat systemic pain is ongoing, it must have been introduced for more than 3 days (according to criteria 3)
* If antidepressant treatment is in progress, it must have been established for over a month for a tricyclic and for more than 15 days for other classes of antidepressants.
* If an anti-epileptic treatment analgesic is in progress, it must have been established for over 15 days.
* Signing of the informed consent form.
* Patient able to respond the self-assessment questionnaires (sufficient understanding assessments, proficiency in French).
* Patient affiliated to an health insurance plan

Exclusion Criteria:

* Allergy to morphine or carboxymethylcellulose or history of intolerance to morphine
* Analgesic at baseline including systemic morphine to greater than 60 mg equivalent dose of morphine treatment
* Fistulated wound
* Heavily exuding wound
* Wound bleeding (spontaneous bleeding)
* Ongoing radiotherapy on chronic wound
* Creatinine > 110 µmol/L, Total bilirubin > 20 µmol/L
* Not communicating patient
* Unable to comply with requirement of the protocol (11 days)
* Patient pregnant or of childbearing age without contraceptive therapy or lactating
* Person deprived of liberty or under guardianship
* Only for pharmacokinetic analysis: analgesics at baseline including morphine or hydromorphone or oxycodone or codeine. Fentanyl is allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2014-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Proportion of patients whose maximum daily consumption in immediate-release oral morphine is less than or equal to 30 mg for the last 72 hours of the study | 11 days
  Proportion of patients whose maximum daily consumption in immediate-release oral morphine is less than or equal to 30 mg (either up to 3 tablets 10 mg per day) for the last 72 hours of the study (day 8 to day 11) and for which the basic treatment is unchanged throughout the duration of the study

SECONDARY OUTCOMES:
Reduction in average daily pain intensity score on a numerical rating scale self assessment, measured on an 11-point between day 1 and day 11 | 11 days
  Reduction in average daily pain intensity score on a numerical rating scale (where 0=no pain and 10=worst possible pain) self assessment, measured on an 11-point between day 1 and day 11. Therefore patients evaluate each morning local pain of the previous 24 hours.
Evaluate the percentage of local pain relief for 24 hours on a rating scale from 0 to 100% | 11 days
Assess and characterize the evolution of local pain on a global impression scale change : Pain related Patient Global Impression of Change (PGIC) and Clinical Global Impression of Change (CGIC) | 11 days
Assess patient satisfaction with treatment of local pain (score 0-4) | 11 days
Evaluate the impact score of local pain on sleep (self-report scale of 0 to 100%) | 11 days
  0% no impact of pain on sleep 100% maximum impact of pain on sleep, inability to sleep
Determine the time (in hours) before using oral immediate-release morphine after application of local treatment | 11 days
Determination of cumulative dose of oral immediate-release morphine (in milligrams) of the 11 days of treatment for relieving painful access of local origin | 11 days
Evaluate systemic and local side effects of analgesic treatment (incidence, severity and location) | 11 days
Evaluate the systemic absorption of topical morphine blood test after the first application | 11 days

CONTACTS AND LOCATIONS:
Overall Officials: Valerie LAURENT, MD, Principal Investigator — Institut Curie - Hôpital René Huguenin; Audrey Hurgon, MD, Study Director — Institut Curie Paris
Locations (5):
- France (5):
  - Hôpital Louis Mourier, Colombes, Île-de-France Region
  - Institut Curie, Paris, Île-de-France Region
  - Hôpital Jean-Jaurès, Paris, Île-de-France Region
  - Groupe Hospitalier Bichat, Paris, Île-de-France Region
  - Institut Curie - Hôpital René Huguenin, Saint-Cloud, Île-de-France Region